CLINICAL TRIAL: NCT00525603
Title: A Phase II Study of Cyclophosphamide, Fludarabine, Alemtuzumab, and Rituximab (CFAR) in High-Risk Previously Untreated Patients With CLL
Brief Title: CFAR Study in Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0269
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Results first posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-01

CONDITIONS: Leukemia; Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CML; Leukemia; Cyclophosphamide; Fludarabine; Alemtuzumab; Rituximab; CFAR
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Alemtuzumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CFAR (Experimental): CFAR = Cyclophosphamide 200 mg/m^2/day 3-5 intravenous (IV) 5-30 minutes, Fludarabine 20 mg/m^2/day 3-5 IV 5-30 minutes, Alemtuzumab 30 mg 1, 3,5 IV 2-4 hours, and Rituximab 375 mg/m^2/day 2 IV 4-6 hours
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Alemtuzumab; Drug: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide — 200 mg/m^2/day 3-5 IV 5-30 minutes
  Other Names: Cytoxan®; Neosar®
Drug: Fludarabine — 20 mg/m^2/day 3-5 IV 5-30 minutes
  Other Names: Fludara®; Fludarabine Phosphate
Drug: Alemtuzumab — 30 mg Days 1, 3, 5 IV 2-4 hours
  Other Names: Campath; Campath-1H
Drug: Rituximab — 375 mg/m^2/day 2 IV 4-6 hours
  Other Names: Rituxan®

SUMMARY:
Primary Objective:

1. Evaluate the ability of Cyclophosphamide, Fludarabine, Alemtuzumab, and Rituximab (CFAR) to increase the proportion of patients with <5% CD5/CD19+ cells in bone marrow to 66% following 3 courses of treatment without significantly increasing the incidence of pneumonia or sepsis compared to a historic group of patients treated with the combination fludarabine, cyclophosphamide, and rituximab (FCR).

Second Objectives:

1. Assess complete remission (CR), nodular partial remission (nPR), and partial remission (PR) rates (overall response) in high-risk, previously untreated patients with CLL treated with CFAR.
2. Evaluate molecular remission in bone marrow by polymerase chain reaction (PCR) for the clonal immunoglobulin heavy chain variable gene in responders treated with CFAR.
3. Assess immune parameters including blood T cell counts and subset distribution and serum immunoglobulin levels pretreatment, during treatment, and post-treatment in patients treated with CFAR.

DETAILED DESCRIPTION:
Fludarabine is a chemotherapy drug that is approved for the treatment of patients with Chronic Lymphocytic Leukemia (CLL). Cyclophosphamide is also a chemotherapy drug that is commonly used to treat patients with CLL. Rituximab and alemtuzumab are special proteins (antibodies) that specifically target and attach to proteins on leukemia cells. These targeted proteins may also be present on normal blood cells. When these antibodies bind to the proteins on leukemia cells, they may help to stop or slow the growth of the disease. The combination of fludarabine, cyclophosphamide, and rituximab has been used in the treatment of previously untreated patients with CLL. The purpose of this study is to see if there is added benefit with the addition of alemtuzumab to this combination.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete physical exam, including routine blood tests (about 3 tablespoons). You may have either a chest x-ray or a computerized tomography (CT) scan if your doctor thinks it is necessary. If you have not had a bone marrow biopsy collected in the past 4 months, you will have a bone marrow sample collected at this time. To collect a bone marrow biopsy, an area of the hip or chest bone is numbed with anaesthetic, and a small amount of bone marrow is withdrawn through a large needle. Women who are able to have children must have a negative blood or urine pregnancy test.

If you are found to be eligible to take part in this study, you may begin treatment. During this study, you will have up to 6 "cycles" of treatment. A cycle is made up of treatment with the study drugs for 5 days in a row, then around 3 and a half weeks (23 days) of no treatment with the study drugs. On Days 1, 3, and 5 of each cycle, you will receive alemtuzumab through a needle in a vein. On Day 2 of each cycle you will receive rituximab through a needle in a vein. Cyclophosphamide and fludarabine will be given separately on Days 3, 4, and 5 of each cycle through a needle in a vein. In addition to the study drugs, you may also be given premedication and fluids by vein to help decrease the risk of side effects. The premedication may include steroids that are used to decrease the risk of side effects from the alemtuzumab and rituximab. They will be given before each dose of the alemtuzumab and rituximab. The infusions for each daily treatment visit should take less than 6 hours. This treatment will be given on an outpatient basis. The combination treatment will be repeated every 4 weeks (1 cycle) for a total of up to 6 cycles.

You will receive acetaminophen (Tylenol) by mouth and diphenhydramine hydrochloride (Benadryl) by mouth or vein 30-60 minutes before each dose of rituximab and alemtuzumab. You will also receive hydrocortisone (a steroid) by vein before the first dose of alemtuzumab of each cycle. These drugs will be used to help decrease the risk of side effects. If side effects occur during a treatment, the doses of the drugs may be adjusted (up or down) until the symptoms are gone. Also, if you experience side effects during treatment, you must stay in the clinic to be observed, for 2 hours after the drug is given.

During the treatment and for 2 months after completion of treatment, you will need to take antibiotics to decrease the risk of developing infection.

Trimethoprim/sulfamethoxazole (Bactrim DS, SMX) is a sulfa-drug, and you will be given this to decrease the risk of a type of pneumonia called PCP pneumonia. If you are allergic to sulfa drugs, a similar antibiotic may be given. You will take Valtrex to decrease the risk of potential virus reactivation, including herpes. If you are allergic to Valtrex, a similar antibiotic may be given. You may receive an antibiotic called valganciclovir (Valcyte) to decrease the risk of another virus called cytomegalovirus. You may also take allopurinol for the first week of the first course of treatment. This will help decrease the risk of kidney damage from rapid destruction of your leukemia cells.

During the Cycle 1 of treatment, you will have blood drawn (about 2 tablespoons) for routine blood tests once a week. Then, these blood tests will be repeated before the start of each additional cycle (every 4 weeks). You will also see your treating doctor and provide a history and have a routine physical exam done before each cycle of treatment.

After 3 cycles of treatment, you will have a physical exam and routine blood tests (about 2 tablespoons). You may also have either an x-ray or a CT scan. You will have another bone marrow sample collected. These tests will be used to see if the disease is responding to treatment. If it is found that the disease is not responding to treatment after the first 3 cycles of therapy, you will be taken off the study, and your doctor will discuss other treatment options with you. If it is found that the disease is responding to treatment, another 3 cycles (12 weeks) of treatment will be given. During these additional 3 cycles of therapy, you will have blood drawn (about 2 tablespoons) once a week for routine blood tests.

After 6 cycles of treatment, you will have a physical exam, around 2 tablespoons of blood drawn for routine blood tests, and a bone marrow aspirate and biopsy to determine if your leukemia is in remission.

If your disease gets worse or you experience any intolerable side effects, you will be taken off the study, and your doctor will discuss other treatment options with you.

Around 3-6 months after you receive your last treatment cycle, you will have a physical exam and routine blood tests (about 2 tablespoons). After that, you will have a physical exam and routine blood tests (about 2 tablespoons) every 6 months for the next 2 years. If the leukemia has gone into remission, you will have a bone marrow aspirate and biopsy at 6 months, 1 year, and 2 years after your last treatment cycle, to make sure it stayed in remission. If your disease returns or if you start a new therapy, you will not need to return for these visits. However, you should inform the study doctor/staff that you are receiving other treatment.

This is an investigational study. All of the drugs used in the study are FDA approved and commercially available. Their use together in this study, however, is experimental. As many as 60 patients will take part in the study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of CLL by immunophenotyping and flow cytometry analysis of blood or bone marrow and be previously untreated.
* All patients must be younger than 70 years and have a serum beta-2 microglobulin of >/= 4.0mg/L.
* All patients with Rai stage III-IV are eligible for treatment on this protocol. - OR - All patients with Rai stage 0-II who meet one or more indication for treatment as defined by the NCI-sponsored Working Group are eligible for treatment on this protocol.
* All patients must have a Zubrod performance status of 0-3.
* All patients must have adequate renal and hepatic function (serum creatinine </= 2mg/dL; total bilirubin </= 2.5mg/dL). Patients with renal or liver dysfunction due to organ infiltration by lymphocytes may be eligible after discussion with the Principle Investigator and appropriate dose adjustment considered.
* Patients may not receive concurrent chemotherapy, radiotherapy, or immunotherapy. Localized radiotherapy to an area not compromising bone marrow function does not apply, nor do hematopoietic growth factors such as erythropoietin, Granulocyte colony-stimulating factor (G-CSF), Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF), etc.
* Patients must not have untreated or uncontrolled life-threatening infection.
* Patients must sign informed consent.

Exclusion Criteria:

Patients older than 70 years.

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Wierda, M.D., Ph.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's internet site — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 6/24/2005 to 6/21/2007. All participants were registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Of the 60 enrolled, 60 eligible participants were included in this study and started study drug.
Groups:
- CFAR: Participants received fludarabine 20 mg/m^2 days 3-5 intravenous (IV), cyclophosphamide 200 mg/m^2 days 3-5 IV, Alemtuzumab 30 mg IV days 1, 3 and 5, and rituximab 375 mg/m^2 IV on day 2 for C1 and 500mg/m^2 IV on day 2 for C2-6.
Period: Overall Study
Arm/Group | CFAR
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CFAR
Number analyzed (Participants) | 60
Age Continuous [Median (Full Range); unit: years] | 60 [42 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 45
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Overall Participant Response
Description: Overall Response: Complete remission (CR), nodular partial remission (nPR), and partial remission (PR) rates (overall response) in high-risk, previously untreated patients with CLL treated with CFAR. National Cancer Institute - Working Group (NCI-WG) response criteria. CR defined as zero nodes, Liver/spleen not palpable, zero symptoms, polymorphonuclear leukocyte (PMN)>1,500/uL, Platelets >100,000uL, Hemoglobin (untransfused) >11.0g/dL, Lymphocytes <4,000/uL and Bone Marrow Aspirate biopsy <30% lymphocytes with no lymphocyte infiltrate; PR defined as nodes >/= 50% decrease,Liver/spleen >/= 50% decrease, symptoms not applicable, PMN >1,500/uL or >50% improvement from baseline, Platelets 100,000uL or >/=50% decrease improvement from baseline, Hemoglobin (untransfused) >11.0g/dL or >50% improvement from baseline, Lymphocytes >50% decrease and Bone Marrow Aspirate biopsy Not Applicable for PR; with nPR defined same as PR but with <30% lymphocytes with residual disease on biopsy.
Time Frame: Evaluated after 3 courses of 4 week therapy (12 weeks)
Population: Sixty participants were analyzed for response. Four participants did not have a response and one participant was not evaluable.
Measure: Number; unit: Participants
Arm/Group | CFAR
Number analyzed (Participants) | 60
Participants
  Complete remission (CR) | 44
  Nodular partial remission (nPR) | 1
  Partial remission (PR) | 10

ADVERSE EVENTS:
Time Frame: 5 years 7 months
Arm/Group | CFAR
Serious Adverse Events (participants affected / at risk) | 11/60
Other Adverse Events (participants affected / at risk) | 52/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CFAR (N=60)
Fever (General disorders) | 5 (5)
Elevated Creatinine (Metabolism and nutrition disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 5 (5)
Syncope (Nervous system disorders) | 1 (1)
Febrile Neutropenia (General disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CFAR (N=60)
Drug Reaction (General disorders) | 44 (44)
Nausea (Gastrointestinal disorders) | 37 (37)
Vomiting (Gastrointestinal disorders) | 13 (13)
Constipation (Gastrointestinal disorders) | 10 (10)
Sinusitis (Infections and infestations) | 6 (6)
Fatigue (General disorders) | 20 (20)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Hypotension (Cardiac disorders) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Urinary Tract Infection (Infections and infestations) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 4 (4)
Chest Pain (General disorders) | 4 (4)
Upper Respiratory Infection (Infections and infestations) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 9 (9)
Infection Other (Infections and infestations) | 5 (5)
Mucositis (Infections and infestations) | 3 (3)
Pain Other (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No